CLINICAL TRIAL: NCT00104065
Title: A Phase II, Multicenter, Randomized, Double-Blind, Placebo-Controlled Trial of the Safety and Efficacy of CG53135-05 Administered Intravenously as a Single Dose for the Prevention of Oral Mucositis in Patients Receiving Autologous Hematopoietic Stem Cell Transplant
Brief Title: Safety and Efficacy of CG53135-05 in the Prevention of Oral Mucositis in Patients Receiving Bone Marrow Transplant
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: CuraGen Corporation (Industry)
Responsible Party: Sponsor
Organization: Celldex Therapeutics (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: C-421; NCT00124592 (obsolete NCT alias)
Record Dates: First submitted 2005-02-22; First posted 2005-02-23 (Estimated); Last update posted 2016-03-15 (Estimated); Status verified 2016-02

CONDITIONS: Stomatitis
Keywords: oral mucositis; oncology - supportive care; mouth diseases
MeSH Terms: conditions — Stomatitis; Mouth Diseases | interventions — FGF20 protein, human

INTERVENTIONS:
Drug: CG53135-05, velafermin

SUMMARY:
CG53135-05, a recombinant human fibroblast growth factor-20 (rhFGF-20) protein, is under investigation for the prevention of oral mucositis. Oral mucositis is a commonly occurring side effect of high-dose chemotherapy in patients undergoing autologous hematopoietic stem cell transplant. The objective of this Phase II trial is to evaluate the safety and efficacy of CG53135-05 when administered as a single dose to patients at risk for developing oral mucositis.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients ages > 18 yrs
* Patients undergoing high dose chemotherapy with or without radiation therapy treatment as conditioning for autologous hematopoietic stem cell transplantation. The conditioning regimens include at least one of the following: high dose melphalan (Mel 200), busulfan, or etoposide, with or without total body irradiation.
* Patients with Karnofsky performance scores > or = 70%
* Informed consent for participation in study

Exclusion Criteria:

* Patients who weigh < 33 kg
* Premenopausal female patients who are pregnant, lactating or are likely to become pregnant
* Patients with active medical conditions that preclude autologous hematopoietic stem cell transplantation
* Patients diagnosed with active acquired immunodeficiency syndrome (AIDS) or Hepatitis B/C
* Patients with known hypersensitivity to recombinant protein therapeutics
* Patients who have taken CG53135-05, palifermin or other investigational drugs in the past 30 days
* Patients who have untreated symptomatic dental infection
* Patients with a history of sensitivity or allergy to E. coli-derived products
* Patients with WHO Grade 3 or 4 oral mucositis (OM)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2005-01; Primary Completion 2005-12 (Actual); Study Completion 2005-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (9):
- United States (9):
  - Research Facility, La Jolla, California
  - Research Facility, Denver, Colorado
  - Research Facility, Miami, Florida
  - Research Facility, Chicago, Illinois
  - Research Facility, Worcester, Massachusetts
  - Research Facility, New York, New York
  - Research Facility, Winston-Salem, North Carolina
  - Research Facility, Cleveland, Ohio
  - Research Facility, Portland, Oregon